CLINICAL TRIAL: NCT06017804
Title: A Comparative Study of Muscle Energy Technique and Foam Roller Self-myofascial Release for Chronic Low Back Pain in Two-wheeler Riders
Brief Title: Muscle Energy Technique and Foam Roller Self Myofascial Release in Two-wheeler Riders With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Collaborators: Manav Rachna International Institute of Research and Studies (MRIIRS) (Unknown)
Responsible Party: Principal Investigator, AMIR IQBAL, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRIIRS/FAHS/PT/2022-23/M-010
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Chronic Low-back Pain
Keywords: Hamstring flexibility; Muscle Energy technique; Self-myofascial release; Foam roller; Dynamic balance; Physical disability; Sit and reach test; Active knee extension

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MET Group (Experimental): Received a muscle energy technique
  Interventions: Other: Muscle energy technique
- SMFR Group (Active Comparator): Received a self-myofascial release technique using a foam roller
  Interventions: Other: Self-myofascial release technique

INTERVENTIONS:
Other: Muscle energy technique — Participants were required to adopt a supine position. MET's post-isometric relaxation method was chosen. The therapist gently flexed the patient's hip until the limitation bar-rier was detected. At this stage, isometric contractions against resistance were applied. After that, the patients were told to resist the movement with only 25% of their strength. Before the leg was released, the contraction was maintained for 7-10 seconds. On exhale, the knee joint was straightened (extended) towards its new barrier, and a stretch was applied and maintained through that barrier for 30 seconds. This procedure was carried out six times.
  Arms: MET Group
Other: Self-myofascial release technique — A foam roller was rolled from the ischial tuberosity to the back of the knee on the side being tested while the participant remained seated in a long sitting position. Individuals were instructed to keep all of their body weight on the leg being evaluated. They spent 30-40 seconds rolling one hamstring at a time in each set (10 times back and forth).
  Arms: SMFR Group

SUMMARY:
Pain in the lower back is a major concern in today's era due to prolonged sitting in two-wheeler riders, mainly due to hamstring tightness. It also creates physical disability and impairment in activities of daily living. This study aimed to compare the efficacy of muscle energy technique (MET) and self-myofascial release (SMFR) using the foam roller on hamstring flexibility, dynamic balance, and physical disability amongst two-wheeler riders with chronic low back pain. Participants were randomized into two intervention groups, MET and SMFR, using the envelope method, with each group having 20 participants. Hamstring flexibility and range of motion for knee extension and the lower back were assessed using the active knee extension test and sit and reach test, the dynamic balance was assessed by the star excursion balance test (SEBT) and physical disability by Roland-Morris Disability Questionnaire, (RMDQ). Measurements were taken at baseline and after 4-week of intervention. The level of significance value was set at 95% (p <0.05).

DETAILED DESCRIPTION:
The present study proved that both SMFR using the foam roller and MET are effective in improving hamstring muscle flexibility, dynamic balance, and physical disability in two-wheeler riders with chronic low back pain. Thus, either of the two techniques can be used for treating bikers with tight hamstrings causing chronic low back pain. Compared to MET, SMFR using foam rollers was found to be more effective in enhancing hamstring flexibility, improving balance, and decreasing disability levels on the RMDQ after 4 weeks. This study will be aware of the necessity of hamstring stretching and balance training among two-wheeler riders for a prolonged duration on a daily basis and take the initiative to improve their hamstring flexibility and balance.

ELIGIBILITY:
Inclusion Criteria:

* Two-wheeler riders of either gender between the ages of 20 and 40 years,
* Who had ridden at least two hours per day for the previous two years,
* Had musculoskeletal pain in the back for the previous three months, and
* Had a 15-20-degree loss of knee extension when hips were held in 90-degree flexion.

Exclusion Criteria:

* Pregnant women,
* Those with a recent spine or lower limb fracture, recent surgery,
* A previous hamstring injury,
* Lumbar and lower limb neurological deficits, or limb length disparity.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Hamstring flexibility | 4 weeks
  Hamstring flexibility was assessed using an active knee extension test (AKET) at baseline and four weeks post-intervention.
Active range of motion | 4 weeks
  Active range of motion was assessed using a sit and reach test (SRT) at baseline and four weeks post-intervention.
Dynamic balance | 4 weeks
  Dynamic balance was assessed using a star excursion balance test (SEBT) at baseline and four weeks post-intervention.
Roland-Morris Disability Questionnaire Scale | 4 weeks
  Roland-Morris Disability Questionnaire (RMDQ) was used assessing the physical disability at baseline and four weeks post-intervention. The RMQ is a 24-item patient-reported outcome measure that inquires about pain-related disability resulting from LBP. Items are scored 0 if left blank or 1 if endorsed, for a total RMQ score ranging from 0 to 24; higher scores represent higher levels of pain-related disability.

CONTACTS AND LOCATIONS:
Overall Officials: AMIR IQBAL, MPT, Study Chair — King Saud University
Locations (1):
- Department of Rehabilitation Sciences, College of applied Medical Science, King Saud University, Riyadh, Saudi Arabia